CLINICAL TRIAL: NCT02903082
Title: Following of Myeloid-derived Suppressor Cells (MDSC) in Severe Sepsis: What Relationship With Systemic Inflammatory Syndrome?
Acronym: MDSC
Status: Terminated | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I16019 (MDSC)
Record Dates: First submitted 2016-09-02; First posted 2016-09-16 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Severe Sepsis; Inflammatory Response Syndrome, Systemic
Keywords: Myeloid-Derivated suppressive cell; Sepsis; Inflammatory Response Syndrome, Systemic
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome | interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residue of blood further to NFS for case
  Bone marrow collected during myelogram routinely performed during hospitalization in ICU
  Blood samples collected routinely as part of a preoperative workup for control
  Bone marrow collected during a myelogram carried out for hematological pathology workup for control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Patient hospitalized in intensive care for sepsis evolving for less than 48 hours with two criteria of systemic inflammatory response syndrome
  Interventions: Biological: Residue of blood further to NFS; Biological: Bone marrow collected during myelogram routinely performed during hospitalization in ICU
- Control: 10 Patients hospitalized for a hematologic pathology workup considered normal by two haematologists and 10 patients hospitalized for a preoperative workup.
  Interventions: Biological: Residue of blood further to preoperative workup; Biological: Bone marrow collected during a myelogram carried out for hematological pathology workup

INTERVENTIONS:
Biological: Residue of blood further to NFS
  Groups: Case
Biological: Residue of blood further to preoperative workup
  Groups: Control
Biological: Bone marrow collected during a myelogram carried out for hematological pathology workup
  Groups: Control
Biological: Bone marrow collected during myelogram routinely performed during hospitalization in ICU
  Groups: Case

SUMMARY:
Sepsis remains a major cause of death in developed countries. A better understanding of the mechanisms involved in the regulation of inflammatory and immune response of patients with severe sepsis is an important step that could open the way for new therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old
* Patient with two criteria of systemic inflammatory response syndrome and one of the four following criteria within 24 hours of hospitalization in ICU:

  * Lactate >4 mmol/L
  * PaO2 / FiO2 <200 in the presence of lung disease as infectious source
  * Vasopressor: adrenaline or noradrenaline ≥0.25 µg/kg/min for at least 6 hours to maintain a systolic blood pressure ≥90 mmHg or mean arterial pressure ≥65 mmHg
  * Thrombocytopenia linked to sepsis with platelet count <100,000 / ml or a decrease ≤50% within 48 hours

Exclusion Criteria:

* Pregnancy
* progressive solid cancer
* HIV infection
* History of blood or inflammatory disease
* long-term immunosuppressive treatment
* Prior episode of Sepsis in the previous month
* Chronic Dialysis Patient
* Patient under guardianship
* Patient not affiliated with a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in intensive care for sepsis evolving for less than 48 hours with two criteria of systemic inflammatory response syndrome
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Peripheral Blood MDSC concentration during ICU hospitalization for Severe Sepsis | Average 30 days - Patients will be followed up until hospital discharge
  Number of patients showing an increase of Myeloid derived suppressive cells from baseline at Day 30.
  Kinetic of Myeloid derived suppressive cells through weekly measures of Absolute Cell Counts (using flow cytometry)

SECONDARY OUTCOMES:
Immuno- inflammatory status | Day 0, Day3, Day 7 and once a week until the intensive care unit discharge
  Pro-inflammatory cytokines determined by flow cytometry
MDSCs presence in the blood and bone marrow. | Day 0
  Concentration of MDSC in the blood determined by flow cytometry
Assessment of MDSC specific gene expressions | Day 0 vs Days 3, 7, 14, 21, 28
  Measurement of MDSC activation by real-time qRT-PCRMDSC cell culture
Assessment of MDSC functional status | Day 0 vs Days 3, 7, 14, 21, 28
  Inhibition of T cell proliferation capacity (co-culture assay in vitro)MDSC cell culture
Mortality | Day 28 and Day 90
  Dead or alive
Incidence of hospital acquired secondary infections at Day 28 | Day 28
  Incidence of hospital acquired secondary infections at Day 28
SOFA score | Day 0, Day3, Day 7 and once a week until the intensive care unit discharge
  Calculating of SOFA score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de LIMOGES, Limoges, France